CLINICAL TRIAL: NCT01651416
Title: An Individually Randomised Trial of Seasonal Malaria Chemoprevention Versus a Long-acting Artemisinin Combination Therapy for the Prevention of Malaria and Anaemia in Children Living in an Area of Extended Seasonal Transmission in Ghana.
Brief Title: Seasonal Malaria Chemoprevention Versus Home Management of Malaria in Children Under 5 Years in Ghana
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Global Health Research, Ghana (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Harry Tagbor, Principal Investigator, Centre for Global Health Research, Ghana
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QA389
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Malaria; Anaemia
Keywords: Home management of malaria; Seasonal malaria chemoprevention
MeSH Terms: conditions — Malaria; Anemia | interventions — Artemether, Lumefantrine Drug Combination; Amodiaquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HMM using short-acting ACT (Active Comparator): Home management of malaria using Artemether-lumefantrine combination (a short-acting ACT) for treatment in children with malaria diagnosed using RDTs
  Interventions: Drug: Artemether-lumefantrine combination
- HMM using short-acting ACT plus SMC (Experimental): Home management of malaria using using Artemether-lumefantrine combination (a short-acting ACT) for treatment in children with malaria diagnosed using RDTs plus seasonal malaria chemoprevention with Amodiaquine plus sulphadoxine-pyrimethamine combination.
  Interventions: Drug: Artemether-lumefantrine combination; Drug: Amodiaquine plus sulphadoxine-pyrimethamine combination
- HMM using a long-acting ACT (Experimental): Home management of malaria using Dihydroartemisinin Piperaquine combination (a long-acting ACT) for treatment in children with malaria diagnosed using RDTs
  Interventions: Drug: Dihydroartemisinin Piperaquine combination

INTERVENTIONS:
Drug: Artemether-lumefantrine combination
  Arms: HMM using short-acting ACT; HMM using short-acting ACT plus SMC
Drug: Dihydroartemisinin Piperaquine combination
  Other Names: Duo-cotecxin
  Arms: HMM using a long-acting ACT
Drug: Amodiaquine plus sulphadoxine-pyrimethamine combination
  Arms: HMM using short-acting ACT plus SMC

SUMMARY:
In areas of Africa where malaria is only a problem during a short rainy season, monthly courses of antimalarial drugs can provide very effective prevention of malaria in children. This approach, called intermittent preventive treatment in children (IPTc) but now known as Seasonal Malaria Chemoprevention (SMC), may also be useful in large areas of Africa where malaria is transmitted for longer each year. It is uncertain if IPTc would be effective, acceptable to communities or sustainable when delivered over a longer period, but this is an important public health question of key interest to policy makers, because in areas with a longer transmission season, the burden of malaria is typically higher than in highly seasonal areas.

Another form of prevention that would be operationally easier for African countries to put into practice would be to treat malaria patients with long-lasting antimalarials, which protect children against further malaria episodes for several weeks. Because malaria disproportionately affects certain high risk children more than others, causing repeated attacks of fever and leading to severe anaemia, long-acting drugs may be a simple and effective way to target limited resources at the individuals who most need protection. This may be particularly beneficial where malaria is a seasonal problem, because repeated malaria attacks will not only be borne by a few unfortunate children, but will also occur close together in time.

The investigators propose a clinical trial to evaluate these two forms of chemoprevention in Kumasi, Ghana, an area with an extended malaria transmission season. Children under 5 years of age currently have access to diagnosis and treatment of malaria via by community based health workers. Children enrolled in the study will receive either the standard community-based diagnosis and treatment, treatment with a longer-acting artemisinin combination therapy (ACT), or standard care plus five monthly courses of seasonal malaria chemoprevention (SMC) during the peak in transmission.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 3-59 months
* Care giver or parent willing to participate and have given informed consent
* Children living in the study area

Exclusion Criteria:

* Children who are unable to take and retain medication
* Children who have a severe or chronic illness
* Children who have a history of serious adverse reaction to the study drugs

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2400 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Incidence of malaria cases | 12 months
  Incidence of malaria cases recorded by the community health workers (CHWs) and at the study health centres. Malaria will be defined as fever or history of fever combined with parasitologically confirmed P. falciparum infection by blood slide. Management of suspected malaria cases reporting to CHWs and health centres will be according to rapid diagnostic test (RDT).

SECONDARY OUTCOMES:
Proportion of children with parasitaemia | 12 months
  Parasitaemia detected by rapid diagnostic test (RDT) and parasitologically confirmation of P. falciparum infection by blood slide..
Proportion of children with anaemia | 12 months
  Anaemia is defined as haemoglobin less than <8 g/dL
Number of referrals | 12 months
  Referrals to hospital and admissions due to malaria and other causes
Incidence of severe illness | 12 months
Incidence of adverse events | 12 months

OTHER OUTCOMES:
Acceptability of seasonal malaria chemoprevention | 2 months
  Acceptability of seasonal malaria chemoprevention through Focus Group Discussions and in-depth interviews

CONTACTS AND LOCATIONS:
Overall Officials: Harry Tagbor, DrPH, Principal Investigator — Kwame Nkrumah University of Science and Technology
Locations (1):
- Ejisu-Juaben Municipality, Kumasi, Ashanti Region, Ghana